CLINICAL TRIAL: NCT01829802
Title: A Pilot Randomized, Open Label Study to Evaluate Efficacy and Safety of the Combination of RAL+ATV/r in Comparison With TDF/FTC+ATV/r in HIV Infected Patients, Who Failed an Initial NNRTI Containing Regimen
Brief Title: RAL+ATV/r in Comparison With TDF/FTC (or 3TC) +ATV/r in HIV Infected Patients
Acronym: ARTE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pedro Cahn (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Pedro Cahn, President, Fundación Huésped
Organization: Fundación Huésped (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FH-14; 50250 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Infection With HIV
Keywords: HIV; Raltegravir; Boosted atazanavir
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir; Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RAL+ATA/r (Experimental): Raltegravir 400 mg BID plus Ritonavir Boosted Atazanavir 300/100 mg QD
  Interventions: Drug: Ritonavir boosted Atazanavir; Drug: Raltegravir
- TDF/FTC (or 3TC) +ATA/r (Active Comparator): TDF/FTC (or 3TC)- Fixed dose combination of Tenofovir 300 mg plus Emtricitabine 200 mg (or Lamivudine 300 mg) QD plus Ritonavir Boosted Atazanavir 300/100 mg QD
  Interventions: Drug: Ritonavir boosted Atazanavir; Drug: TDF/FTC (or 3TC)

INTERVENTIONS:
Drug: Ritonavir boosted Atazanavir — Ritonavir boosted Atazanavir 300/100 mg QD in combination with other drugs
  Other Names: Reyataz; Norvir
Drug: Raltegravir — Raltegravir 400 BID in combination with Ritonavir boosted Atazanavir 300/100 mg QD during 48 weeks
  Other Names: Isentress
  Arms: RAL+ATA/r
Drug: TDF/FTC (or 3TC) — Fixed dose combination of Tenofovir 300 mg/Emtricitabine 200 mg or Tenofovir 300 mg/Lamivudine 300 mg plus Ritonavir Boosted Atazanavir 300/100mg given once a day
  Other Names: Truvada; TDF-FTC; TDF-3TC; Mivuten
  Arms: TDF/FTC (or 3TC) +ATA/r

SUMMARY:
The purpose of this pilot study is to assess the efficacy and safety of the combination of RAL+ATV/r in comparison with TDF/FTC+ATV/r in HIV-1 infected patients presenting virologic failure and PI and TDF naïve.

DETAILED DESCRIPTION:
Overall Study Design and Plan: Description

This is a pilot, randomized, open-label study. All the participants will be assigned to receive RAL+ATV/r or TDF/FTC+ATV/r. Patients will be evaluated at screening, randomization (day 0), and on weeks 4, 8, 12, 24, 36 and 48.

At the screening visit, subjects must be willing and able to give written (signed and dated) informed consent prior to any study specific procedures. They will receive a unique screening number and will undergo the study procedures associated with the screening visit. The investigator will evaluate whether the subject meets all eligibility criteria specified and record the details of the informed consent process and the results of this assessment in the subject's medical records. Two forms of the ICF will be signed, one for the subject and the other to file at the site.

At baseline visit, enrollment criteria will be reviewed and subjects who meet all of them will undergo study procedures. Subjects will receive instructions about study medications and dosing schedule. Subjects should start study medication within 24 hours of the baseline visit. Subjects will return to the investigator´s site for study visits and procedures. Subjects who prematurely discontinue the study must return for a discontinuation visit and undergo the study procedures identified for the discontinuation visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject ≥18 years of age.
* Documented HIV-1 infection defined as a positive ELISA plus a confirmatory Western Blot; or a plasma HIV-1 RNA ≥10,000 copies/mL ever documented.
* Patients who have failed their initial treatment containing NNRTI(s) + 2NRTI(s) combination therapy, according to virological criteria defined by two consecutive (at least 7 days apart) HIV-1 RNA results ≥500 copies/mL. Subject must be on stable HAART for at least the last 4 weeks.
* No prior or current exposure to HIV-1 protease inhibitors and/or HIV-1 integrase inhibitors.
* Subject must have susceptibility to ATV/r and TDF, as resulted by resistance testing at screening. RAL sensitivity is not required for patients never exposed to this drug in the country.
* Subject has voluntarily signed ICF.
* Subject can comply with protocol requirements.
* Subject's general medical condition, in the investigator's opinion, does not interfere with assessments and completion of the trial.
* Subject agrees not to take any medication during the study, including over the counter medicines or herbal preparations, without the approval of the trial physician.
* If female, is not breastfeeding or pregnant.
* If female, subject must be either postmenopausal for at least one year, surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or she must use 2 different methods of birth control including, at least, one barrier method, that are acceptable to both the subject and investigator, and willing to continue their use for at least 30 days after the end of the treatment period.
* Subjects must have a life-expectancy of more than 1 year.

Exclusion Criteria:

* Patient has a current (active) diagnosis of acute hepatitis due to any cause OR chronic hepatitis B and/or C WITH aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN) AND/OR is likely to require hepatitis treatment in the next year.
* Active hepatitis B infection (positive HBsAg), regardless of stage of infection.
* Subject has a currently active AIDS defining illness (Category C conditions according to the CDC Classification System for HIV infection 1993) in the last 30 days.
* Subjects with a laboratory abnormality Grade 3 or 4 with the following exceptions: pancreatic amylase, cholesterol, triglycerides, gamma glutamyl transpeptidase.
* Screening laboratory analysis show any of the following abnormal results:

  * Hemoglobin <8.0 g/dL
  * Absolute neutrophil count <750 cells/µL
  * Platelet count <50,000 mm3
  * Creatinine >1.5 x ULN
* Any condition that, in the investigators opinion, could compromise the subject's safety or adherence to the trial protocol.
* The use of any study agent within 30 days prior to screening.
* Use of immunosuppressive drugs, cytokines inhibitors or other cytokines in the previous year.
* Any other condition (including, without limitation, the use of alcohol or drugs) that in the investigator's opinion may compromise the safety of the patient or his/her adherence to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV-1 RNA below the limit of detection (<50 copies/mL)in an intention to treat (exposed) analysis. | 48 weeks
Proportion of subjects with SAEs and proportion with AEs leading to discontinuation. | Through week 48

SECONDARY OUTCOMES:
Change from baseline on viral load | 24 and 48 weeks
Change from baseline in lipid profile and renal function | Through 48 weeks
Change from baseline in inflammation markers | 24 and 48 weeks

OTHER OUTCOMES:
Number and type of resistance mutations in case of virologic failure | Through 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Cahn, MD, Principal Investigator — Fundación Huésped
Locations (2):
- Argentina (2):
  - Fundacion Huesped, Buenos Aires, Buenos Aires
  - Dra Luna Norma, Córdoba, Córdoba Province

IPD SHARING:
Plan to Share IPD: Undecided